CLINICAL TRIAL: NCT02174419
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel, 3-Arm Study of the Safety and Anti-Pruritic Efficacy of Nalbuphine HCl ER Tablets in Prurigo Nodularis Patients
Brief Title: Study of Nalbuphine HCl ER Tablets in Patients With Prurigo Nodularis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR03; 2013-005627-17 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Prurigo Nodularis; Nodularis Prurigo; Prurigo; Pruritus
Keywords: Itch; Chronic Itch; nalbuphine
MeSH Terms: conditions — Prurigo; Pruritus | interventions — BID protein, human; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- nalbuphine HCl ER 90mg (Experimental): nalbuphine HCl ER tablets 90 mg BID
  Interventions: Drug: nalbuphine HCl ER tablets 90 mg BID
- nalbuphine HCl ER 180 mg (Experimental): nalbuphine HCl ER tablets 180 mg BID
  Interventions: Drug: nalbuphine HCl ER tablets 180 mg BID
- Sugar pill (Placebo Comparator): Placebo tablets BID
  Interventions: Drug: Placebo tablets BID

INTERVENTIONS:
Drug: nalbuphine HCl ER tablets 90 mg BID — nalbuphine HCl ER tablets 90 mg BID administered for 8 weeks
  Other Names: nalbuphine ER
  Arms: nalbuphine HCl ER 90mg
Drug: nalbuphine HCl ER tablets 180 mg BID — nalbuphine HCl ER tablets 180 mg BID administered for 8 weeks
  Other Names: nalbuphine ER
  Arms: nalbuphine HCl ER 180 mg
Drug: Placebo tablets BID — Placebo tablets BID administered for 10 weeks
  Other Names: sugar pill
  Arms: Sugar pill

SUMMARY:
The primary objectives of the study are to evaluate the effects of two doses of nalbuphine HCl ER tablets on the change from baseline in the worst itch Numerical Rating Scale (NRS) in patients with prurigo nodularis and to evaluate the safety and tolerability in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Subject suffering from generalized prurigo nodularis
* Have demonstrated pruritus intensity during screening
* Male or female who are at least 18 years old at the time of consent

Exclusion Criteria:

* Subject has chronic pruritus resulting from other conditions
* Subject has a history of substance abuse within the past year
* Subject has a known drug allergy to opioids
* Subject is a pregnant or lactating female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (4):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
- University of Münster, Münster, Germany
- Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw, Lower Silesian Voivodeship, Poland

REFERENCES:
- [Derived] Eudy-Byrne R, Riggs M, Hawi A, Sciascia T, Rohatagi S. A population pharmacokinetic-pharmacodynamic model evaluating efficacy of nalbuphine extended-release in patients with prurigo nodularis. Br J Clin Pharmacol. 2023 Jul;89(7):2088-2101. doi: 10.1111/bcp.15663. Epub 2023 Feb 9. PMID 36680419
- [Derived] Stander S, Zeidler C, Pereira M, Szepietowski JC, McLeod L, Qin S, Williams N, Sciascia T, Augustin M. Worst itch numerical rating scale for prurigo nodularis: a psychometric evaluation. J Eur Acad Dermatol Venereol. 2022 Apr;36(4):573-581. doi: 10.1111/jdv.17870. Epub 2022 Feb 14. PMID 34908192
- [Derived] Weisshaar E, Szepietowski JC, Bernhard JD, Hait H, Legat FJ, Nattkemper L, Reich A, Sadoghi B, Sciascia TR, Zeidler C, Yosipovitch G, Stander S. Efficacy and safety of oral nalbuphine extended release in prurigo nodularis: results of a phase 2 randomized controlled trial with an open-label extension phase. J Eur Acad Dermatol Venereol. 2022 Mar;36(3):453-461. doi: 10.1111/jdv.17816. Epub 2021 Dec 1. PMID 34780095

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nalbuphine HCl ER 90mg | Nalbuphine HCl ER 180 mg | Sugar Pill
Started | 22 | 18 | 22
Completed | 18 | 12 | 20
Not Completed | 4 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nalbuphine HCl ER 90mg | Nalbuphine HCl ER 180 mg | Sugar Pill | Total
Number analyzed (Participants) | 22 | 18 | 22 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (8.6) | 49.1 (16.3) | 53.3 (16.7) | 52.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 12 | 34
  Male | 10 | 8 | 10 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 18 | 22 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 20 | 15 | 19 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 6 | 15
  Europe | 17 | 14 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Evaluation Visit (Week 10) in Itch on the 0-10 Numerical Rating Scale
Description: The number of subjects who reported at least a 30% reduction from baseline to Week 10, expressed as a percentage of subjects in the particular arm/group who were evaluated,
Time Frame: Baseline, Week 10
Measure: Number; unit: percentage of subjects
Arm/Group | Nalbuphine HCl ER 90mg | Nalbuphine HCl ER 180 mg | Sugar Pill
Number analyzed (Participants) | 22 | 18 | 22
percentage of subjects | 27.3 | 44.4 | 36.4

2. Secondary Outcome: Change From Baseline to the Evaluation Visit (Week 10) in the Mean Itch on the 0-10 Numerical Rating Scale
Time Frame: Baseline, Week 10
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change From Baseline to the Evaluation Visit (Week 10) in the Verbal Rating Scale
Time Frame: Baseline, Week 10
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Nalbuphine HCl ER 90mg | Nalbuphine HCl ER 180 mg | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/18 | 1/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nalbuphine HCl ER 90mg (N=22) | Nalbuphine HCl ER 180 mg (N=18) | Sugar Pill (N=22)
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No